CLINICAL TRIAL: NCT00690872
Title: Phase II Trial Evaluating Efficacy of a Strategy Employing Combination Gemcitabine and Carboplatin Chemotherapy Followed by EBV-Specific Cytotoxic T-Lymphocytes in Patients With Metastatic or Locally Recurrent EBV-Positive Nasopharyngeal Carcinoma
Brief Title: Gemcitabine and Carboplatin Followed By Laboratory-Treated T Lymphocytes in Treating Patients With Metastatic or Locally Recurrent Epstein-Barr Virus-Positive Nasopharyngeal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000577971; SINGAPORE-07-27-NPC
Record Dates: First submitted 2008-06-04; First posted 2008-06-05 (Estimated); Last update posted 2009-06-29 (Estimated); Status verified 2009-06

CONDITIONS: Head and Neck Cancer
Keywords: recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Carboplatin; Gemcitabine; Polymerase Chain Reaction; Flow Cytometry; Immunoenzyme Techniques

INTERVENTIONS:
Biological: autologous Epstein-Barr virus-specific cytotoxic T lymphocytes
Drug: carboplatin
Drug: gemcitabine hydrochloride
Genetic: polymerase chain reaction
Other: fluorescence activated cell sorting
Other: immunoenzyme technique

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving an infusion of a person's T lymphocytes that have been treated in the laboratory may help the body build an effective immune response to kill tumor cells. Giving combination chemotherapy together with laboratory-treated T lymphocytes may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine and carboplatin together with laboratory-treated T lymphocytes works in treating patients with metastatic or locally recurrent Epstein-Barr virus-positive nasopharyngeal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine progression-free survival (PFS 1) of patients with metastatic or locally recurrent Epstein-Barr virus (EBV)-positive nasopharyngeal carcinoma treated with gemcitabine hydrochloride and carboplatin followed EBV-specific cytotoxic T-lymphocytes (CTL).

Secondary

* To determine progression-free survival (PFS 2) of these patients during the immunotherapy portion of this study.
* To determine the clinical benefit rate of EBV-specific CTL in these patients.
* To determine the tolerability of EBV-specific CTL therapy in these patients.
* To demonstrate persistence of EBV-specific immune response in these patients.

OUTLINE: Patients undergo collection of peripheral blood mononuclear cells (PBMC) from which T cells are purified, co-cultured with irradiated autologous Epstein-Barr virus (EBV)-specific cytotoxic T-lymphocytes (CTLs), and expanded in vitro for the establishment of cytotoxic T-cell lines.

* Chemotherapy: Patients receive gemcitabine hydrochloride IV over 30 minutes and carboplatin IV over 60 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. After completion of course 2, patients undergo evaluation for response. Patients with progressive disease proceed directly to induction immunotherapy. Patients with stable disease (SD), partial response (PR), or complete response (CR) receive 2 additional courses of chemotherapy and then proceed to induction immunotherapy.
* Induction immunotherapy: Beginning 14-28 days after the completion of chemotherapy, patients receive EBV-specific CTLs IV over 1-10 minutes on days 1 and 14. Six weeks after the second infusion, patients undergo evaluation for response. Patients who demonstrate clinical benefit (i.e., CR, PR, SD) to induction immunotherapy proceed to maintenance immunotherapy.
* Maintenance immunotherapy: Patients receive EBV-specific CTLs IV over 1-10 minutes. Treatment repeats every 1-3 months for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection at baseline and prior to each course of induction immunotherapy and maintenance immunotherapy. Samples are analyzed for EBV CTL frequency by immune function assays (i.e., tetramer analysis, enzyme-linked immunospot, and cytotoxic T-lymphocyte precursor assays); for specificity of response by cytotoxicity assays (in patients for whom the appropriate reagents are available); and for evaluation of EBV DNA by polymerase chain reaction. In addition, T-cells are isolated from blood samples for fluorescence-activated cell sorter analysis and for extraction of RNA.

After completion of study therapy, patients are followed at least every 2 months until disease progression.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven nasopharyngeal carcinoma (NPC)

  * WHO type 2/3 disease
  * Metastatic or locally recurrent disease
* Epstein-Barr virus (EBV)-positive disease as confirmed by in situ hybridization assay or PCR amplification for EBV-encoded RNA expression
* Radiologically measurable disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* ANC > 1,200/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8 g/dL
* Bilirubin < 2 times upper limit of normal (ULN)
* AST and ALT < 3 times ULN
* Creatinine clearance ≥ 40 mL/min
* Corrected calcium normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent severe illness, including any of the following:

  * Chronic obstructive pulmonary disease
  * Ischemic heart disease
  * Active congestive cardiac failure
  * Active angina pectoris
  * Uncontrolled arrhythmia
  * Uncontrolled hypertension
* No concurrent severe infections
* HIV negative

PRIOR CONCURRENT THERAPY:

* No more than one line of prior chemotherapy for metastatic disease
* No prior gemcitabine hydrochloride
* Prior platinum agents allowed
* At least 1 month since prior investigational therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-07; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Median progression-free survival (PFS 1), defined as the time from study enrollment to the time of radiological disease progression or death from any cause

SECONDARY OUTCOMES:
Median PFS 2, defined as the time from the start of induction immunotherapy to radiological disease progression or death from any cause
Response rate, defined as the proportion of patients who achieve a complete response (CR) or partial response (PR) after 4 courses of chemotherapy and the proportion of patients who achieve a further response after immunotherapy
Clinical benefit rate of immunotherapy, defined as the proportion of patients who achieve CR, PR, or stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Toh Han Chong, MD, MBBS, MRCP, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre - Singapore, Singapore, Singapore